CLINICAL TRIAL: NCT02717260
Title: Inhibition Control Modulation by Transcranial Random Noise Stimulation (tRNS ) on the Prefrontal Cortex Measured by Change in Go no Test
Brief Title: Inhibition Transcranial Random Noise Stimulation
Acronym: inhibistim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Principal Investigator, HAESEBAERT, MD PhD, Hôpital le Vinatier
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-A01554-45
Record Dates: First submitted 2016-01-28; First posted 2016-03-23 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Impulsive Behavior; Inhibition
MeSH Terms: conditions — Impulsive Behavior; Inhibition, Psychological | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sham transcranial noise stimulation (Sham Comparator): subjects are stimulated 3 times with sham transcranial random noise stimulation (tRNS) (Starstim) with a 30 seconds offset
  Interventions: Device: transcranial random noise stimulation (tRNS) (Starstim)
- 1 Active transcranial random noise stimulation (Active Comparator): subjects are stimulated 1 time with active transcranial random noise stimulation (tRNS) (Starstim) at 2mA with a oscillatory frequency between 100 and 500 Hz during 20 minutes and 2 times with sham tRNS
  Interventions: Device: transcranial random noise stimulation (tRNS) (Starstim)
- 3 Active transcranial random noise stimulation (Active Comparator): subjects are stimulated 3 times with active transcranial random noise stimulation (tRNS) (Starstim) at 2mA with a oscillatory frequency between 100 and 500 Hz during 20 minutes
  Interventions: Device: transcranial random noise stimulation (tRNS) (Starstim)

INTERVENTIONS:
Device: transcranial random noise stimulation (tRNS) (Starstim) — subjects are stimulated 3 times in a day by transcranial random noise stimulation (tRNS) (Starstim). each 20 minutes stimulation are separated by a period of at least 30 minutes. before and after each stimulation, inhibition is evaluated by cognitive tests: go nogo test, stroop test, Hayling test and by the BIS 10 scale. During the stimulation, subjects compleat the STAXI and STAI scales. Cognitive tests are repeated 24 hours and 8 days after the stimulation to evaluate duration of the effect. Possible side effects will be notified throughout the protocol.

SUMMARY:
Inhibition control deficits is a major risk factor in the transition to the act in suicidal patients. Neuroimaging studies have shown that this failure was associated with hypoactivity in the prefrontal cortex (PFC), a brain area involved in the control of impulsivity. It was recently shown that a noninvasive brain stimulation session applied on the PFC reduces transiently impulsivity in healthy volunteers. Noninvasive brain stimulation modulates the activity and connectivity of neural network connected to the stimulation site. The investigators assume that a repetition of noninvasive brain stimulation sessions on the PFC will allow a more intense and longer lasting effect on impulsivity and cognitive control in healthy volunteers compared to a single session and to placebo stimulation. The investigators assume that this behavioral change will be accompanied by a change in brain activity measured by resting EEG for the patients in the active group. A more intense and longer lasting effect is an essential step to transfer these results to patient populations.

The main objective is to study the effect of bilateral stimulation of the PFC by transcranial random noise stimulation (tRNS) on the inhibition control measured by the cognitive motor inhibition capacity (Go NoGo test). The secondary objectives are to study the effect of tRNS on verbal inhibition (measured with the Hayling test); on anxiety (measured with the State-trait anxiety inventory (STAI)),on angry (measured with the State-trait anger expression inventory (STAXI)) on verbal and nonverbal inhibition (measured by the Stroop test), on impulsive behavior (measured by the Barrat impulsiveness scale (BIS 10)) and on the neuronal electrical activity measured by EEG.

DETAILED DESCRIPTION:
Subjects are stimulated 3 times in a day. Each 20 minutes stimulation are separated by a period of at least 30 minutes. Before and after each stimulation, inhibition is evaluated by cognitive tests (Go Nogo test, Stroop test, Hayling test) and by the BIS 10 scale. During the stimulation, subjects compleat the STAXI and STAI scales. Cognitive tests are repeated 24 hours and 8 days after the stimulation to evaluate duration of the effect. Possible side effects will be notified throughout the protocol.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45 years

Exclusion Criteria:

* inability to give consent
* Under 18 years
* over 45 years
* pregnant women
* nursing mothers
* History of neurological or psychiatric disorders and personality disorders in Cluster impulsivity (cluster B) according to Diagnostic and Statistical Manual (DSM) IV
* french National Adult Reading Test (fNART): score below the 5th percentile
* Contraindications to the practice of transcranial brain stimulation as international safety recommendations (Rossi et al., 2009)
* Processing or recent psychotropic

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

PRIMARY OUTCOMES:
Change in go no go test | 15 minutes after the stimulation
  errors and reaction times

SECONDARY OUTCOMES:
Change in Stroop test | 15 minutes after the stimulation
  errors and reaction times
Change in Hayling test | 15 minutes after the stimulation
  errors and reaction times
Change in BIS 10 | 24 hours and 8 days after stimulations
  motor impulsivity, cognitive impulsivity, non planning impulsivity
Change in STAXI | 24 hours and 8 days after stimulations
  score
Change in STAI | 24 hours and 8 days after stimulations
  score
Change in EEG | 24 hours and 8 days after stimulations
occurrence of adverse effects | 8 days after stimulations

CONTACTS AND LOCATIONS:
Overall Officials: HAESEBAERT Frederic, MD PhD, Principal Investigator — HOPITAL VINATIER
Locations (1):
- Ch Le Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No